CLINICAL TRIAL: NCT06299371
Title: A Prospective, Single-arm Study of Adebrelimab in Combination With Paclitaxel for Injection (Albumin Bound) and Platinum Chemotherapy as Neoadjuvant Therapy in Resectable Non-Small Cell Lung Cancer (NSCLC) Harboring Driver Gene Mutations
Brief Title: Adebrelimab Plus Chemotherapy as Neoadjuvant Therapy in Resectable NSCLC Harboring Driver Gene Mutations
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hongxu Liu, Chief Physician, Liaoning Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-NSCLC-II-033
Record Dates: First submitted 2024-02-19; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Injections; 130-nm albumin-bound paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant immuno-chemotherapy (Experimental): Adebrelimab plus paclitaxel for injection (albumin bound) and platinum chemotherapy
  Interventions: Drug: Adebrelimab; Drug: paclitaxel for injection (albumin bound); Drug: Cisplatin or Carboplatin

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab IV
  Other Names: SHR-1316
Drug: paclitaxel for injection (albumin bound) — paclitaxel for injection (albumin bound) IV
  Other Names: Nab-paclitaxel
Drug: Cisplatin or Carboplatin — Cisplatin or Carboplatin IV

SUMMARY:
This is a prospective, single-arm study to investigate the efficacy and safety of Adebrelimab in combination with paclitaxel for injection (albumin bound) and platinum chemotherapy as neoadjuvant therapy in resectable non-small cell lung cancer harboring driver gene mutations

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Resectable non-small cell lung cancer harboring driver gene mutations.
* At least one measurable disease based on Response Evaluation Criteria in Solid Tumors 1.1.
* Have adequate organ function.
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication；Females should not be breastfeeding；Female subjects of childbearing potential as well as males sexually active with women of childbearing potential must be willing to use an adequate method of contraception.
* Voluntarily comply with the treatment protocol.

Exclusion Criteria:

* Previously treated with any anti-tumor therapy;
* Subject with known autoimmune disease
* Subject with known history of testing positive for human immunodeficiency virus (HIV) or known to have acquired immunodeficiency syndrome (AIDS), subject has known active hepatitis B or C.
* Presence of third space effusion that cannot be controlled by drainage or other means (e.g., excessive pleural fluid and ascites).
* Subject with severe liver and kidney dysfunction.
* Subjects who need to use corticosteroids (>10 mg/day prednisone or equivalent dose of similar drugs) or other immunosuppressive therapy for systematic treatment within 14 days before the first administration of the study
* Subject with previous malignancies within 5 years, except for cured in situ cancer.
* Subject with previous or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-induced pneumonia and severe damage to lung function.
* Subject with uncontrolled hypertension.
* Prior organ transplantation including allogenic stem-cell transplantation.
* Known hypersensitivity to the study drug or any of its excipients.
* Other situations that the investigator considers unsuitable for the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | at 12 months
  pCR rate, the proportion of patients achieved pathologic complete response (lung and lymph node without tumor residual assessed by pathology review)

SECONDARY OUTCOMES:
Major pathologic response rate | 12 months
  MPR rate, the proportion of patients achieved pathologic complete response (lung and lymph node ≤10% tumor residual assessed by pathology review)
R0 rate | 12 months
  the proportion of patients achieved R0(No residue under the microscope after resection)
Event Free Survival | up to 5 years
  EFS, the time length from the first dose to any prescriptive events
Overall Survival | up to 5 years
  OS, the time length from the date of the first dose to the date of death.
Objective response rate | 12 months
  ORR, the proportion of patients achieved complete or partial response
Adverse Events | up to 5 years
  AEs

IPD SHARING:
Plan to Share IPD: No